CLINICAL TRIAL: NCT01038336
Title: Hearing Loss Prevention for Veterans
Acronym: HLPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C7214-R; 11-1408 (Other Grant/Funding Number: VA RR&D); 02383 (Other: Portland VAMC IRB committee); 05-2409 (Other: Portland VAMC IRB committee)
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Hearing Loss, Noise-Induced
Keywords: Hearing Loss - Noise-Induced; Prevention; Computer-assisted instruction
MeSH Terms: conditions — Hearing Loss, Noise-Induced

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Multimedia HLPP (Experimental): Multimedia Hearing Loss Prevention Program (HLPP)
  Interventions: Behavioral: Multimedia Hearing Loss Prevention Program
- Hearing Conservation Brochure (Active Comparator): Hearing Conservation Brochure (HCB)
  Interventions: Behavioral: Hearing Conservation Brochure
- Standard-of-Care (No Intervention): Standard-of-Care (SoC)

INTERVENTIONS:
Behavioral: Multimedia Hearing Loss Prevention Program — Interactive, multimedia, computer-based HLPP that provides hands-on education and training about hearing loss, tinnitus, hearing protection, and general hearing health care for Veterans.
  Arms: Multimedia HLPP
Behavioral: Hearing Conservation Brochure — Hearing Conservation brochure provides knowledge-based information similar to that of the multimedia HLPP, but in written form.
  Arms: Hearing Conservation Brochure

SUMMARY:
Hearing loss is the most prevalent service-connected disability in the VA. It causes communication difficulties, which contribute to isolation, frustration and depression. A major cause of hearing loss is from exposure to high levels of sound, and is referred to as Noise Induced Hearing Loss (NIHL). Veterans have inevitably been exposed to high levels of sound during military service, and even though they may not yet have NIHL, their ears have been damaged. Continued noise exposure in civilian life will result in NIHL. However, it can easily be prevented by avoiding noise or using hearing protection. Most people are unaware that noise damages hearing, and even when they are, they do not use hearing protection. In this study we will use a randomized controlled trial to evaluate the short- and long-term effectiveness of two forms of education about NIHL that we have developed for Veterans. One is a computerized program; the other is a Hearing Conservation Brochure

DETAILED DESCRIPTION:
Hearing loss and tinnitus are the two most prevalent service-connected disabilities in the VA system for Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans, and Veterans from World War II, Korea, Vietnam, the Gulf War and during Peacetime. Costs associated with health care utilization, provision of hearing aids, rehabilitation services and reduced productivity for Veterans with hearing loss are substantial, and continue to increase. On a personal level, hearing loss results in communication difficulties, and often contributes to social isolation, frustration and depression. A major cause of hearing impairment is cochlear damage from exposure to high levels of sound. The longer the period of exposure and the more intense the sound pressure level, the greater is the damage that occurs. The damage from noise exposure is cumulative over time, and exacerbates the effects of aging. Veterans, who have been exposed to high levels of sound in the military are therefore highly vulnerable to damage in civilian life, thus they must protect their ears from further noise to avoid hearing loss as they age. Unfortunately, most people are unaware of the damage noise can do to the auditory system, and even when they are aware, few choose to use hearing protection. It is therefore critical to educate Veterans about the dangers of noise exposure and the simple actions that can be taken to protect hearing.

Our long-range goal is to disseminate an effective hearing loss prevention education program that will help to reduce the prevalence and associated costs of noise induced hearing loss in the Veteran population. Ultimately it is our intention to make the program available to all Veterans, military personnel and other members of the public.

We have developed two forms of intervention to educate Veterans about hearing conservation. One is a computerized multimedia interactive program; the other is a printed Hearing Conservation Brochure. Both provide information about hearing, the damage noise can do to the auditory system, the impact hearing loss has on communication, and the use of hearing protection. In this study we will use a randomized controlled trial to evaluate the effectiveness of these two forms of intervention at changing knowledge, attitudes and behaviors toward hearing conservation. Effectiveness will be examined in three ways through assessment of: (1) actual behavioral changes, as evidenced by decreased daily noise exposure as measured with noise dosimetry; (2) reported behavioral changes, as evidenced by decreased daily noise exposure assessed using a real-time log of daily activities and use of hearing protection; and (3) increased knowledge, healthier attitudes and improved intended and actual behavior towards hearing protection, as assessed with a self-report questionnaire. Outcomes will be measured at baseline, immediately following the intervention and six month post-intervention.

There are many challenges facing military personnel as they reintegrate into society after leaving military service. Reducing their risk of acquiring noise induced hearing loss and the associated problems with communication, will help to make this transition less difficult and traumatic. This study will provide important information about the relative effectiveness of two different forms of hearing conservation education. In the long term it has the potential to reduce the prevalence and associated costs of hearing loss and tinnitus among Veterans, and will demonstrate that prevention of hearing loss can reduce the need for long-term rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study all participants will:

* be aged 55 years or less with no exclusions based on ethnicity or gender. The maximum age of 55 years has been selected because hearing conservation programs have the potential to be most effective for younger individuals.
* not use hearing aids
* have cognitive abilities sufficient to participate in the study, as determined by an age/and educationally appropriate score on the Mini Mental State Exam (MMSE).
* ability to read and comprehend the study interventions (HLPP and Hearing conservation brochure) as reflected by a Broad Reading Score of Grade 5 or above on the Woodcock-Johnson III Tests of Achievement Letter-Word Identification, Reading Fluency and Passage Comprehension subtests.
* no known neurological, psychiatric or physical disorders, or co-morbid diseases that would prevent completion of the study as determined by chart review.
* adequate vision to participate in the study as determined with the Smith-Kettlewell Institute Low Luminance (SKILL) Card. Participants will be required to have best corrected vision of 20/63 (mild vision loss) or better.
* openness to using a wearable noise dosimeter and to logging daily activities using a personal digital assistant for three periods of seven days each, as determined by agreement to participate in the study.

Exclusion Criteria:

Individuals will not participate in the study if:

* they are age >55 years.
* wear hearing aids
* score less than the age- and educational-based norms on the MMSE.
* have a Broad Reading score on the Woodcock-Johnson III Tests of Achievement of less than Grade 5.
* have neurological, psychiatric or physical disorders, or co-morbid diseases that would prevent completion of the study.
* have corrected vision poorer than a Snellen equivalent of 20/63.
* be unwilling to use a wearable noise dosimeter and to logging daily activities using a personal digital assistant for three periods of seven days each.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2011-05; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle H Saunders, Principal Investigator — VA Medical Center, Portland
Locations (1):
- VA Medical Center, Portland, Portland, Oregon, United States

REFERENCES:
- [Background] Saunders GH, Griest SE. Hearing loss in veterans and the need for hearing loss prevention programs. Noise Health. 2009 Jan-Mar;11(42):14-21. doi: 10.4103/1463-1741.45308. PMID 19265249
- [Result] Folmer RL, Saunders GH, Dann SM, Griest SE, Porsov E, Fausti SA, Leek MR. Guest editorial: Computer-based hearing loss prevention education program for Veterans and military personnel. J Rehabil Res Dev. 2012;49(4):vii-xvi. doi: 10.1682/jrrd.2012.02.0028. No abstract available. PMID 22773265
- [Result] Saunders GH, Dann SM, Griest SE, Frederick MT. Development and evaluation of a questionnaire to assess knowledge, attitudes, and behaviors towards hearing loss prevention. Int J Audiol. 2014 Apr;53(4):209-18. doi: 10.3109/14992027.2013.860487. Epub 2014 Jan 27. PMID 24467444

RESULTS

PARTICIPANT FLOW:
Groups:
- Multimedia Hearing Loss Prevention Program: Multimedia Hearing Loss Prevention Program (HLPP):
  Multimedia HLPP is an interactive, multimedia, computer-based HLPP that provides hands-on education and training about hearing loss, tinnitus, hearing protection, and general hearing health care for Veterans.
- Hearing Conservation Brochure: Hearing Conservation Brochure (HCB)
  The Hearing Conservation brochure provides knowledge-based information similar to that of the multimedia HLPP, but in written form.
- Standard-of-Care: Standard-of-Care (SoC): SoC amounts to no intervention, however protocol allows participants to independently seek information about hearing loss prevention if they want to..
Period: Overall Study
Arm/Group | Multimedia Hearing Loss Prevention Program | Hearing Conservation Brochure | Standard-of-Care
Started | 43 | 42 | 44
Completed | 43 | 42 | 44
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Multimedia Hearing Loss Prevention Program: Multimedia Hearing Loss Prevention Program (HLPP)
  The multimedia HLPP is an interactive, multimedia, computer-based HLPP that provides hands-on education and training about hearing loss, tinnitus, hearing protection, and general hearing health care for Veterans.
- Hearing Conservation Brochure: Hearing Conservation Brochure (HCB)
  Hearing Conservation brochure: The Hearing Conservation brochure provides knowledge-based information similar to that of the multimedia HLPP, but in written form.
- Total: Total of all reporting groups
Arm/Group | Multimedia Hearing Loss Prevention Program | Hearing Conservation Brochure | Standard-of-Care | Total
Number analyzed (Participants) | 43 | 42 | 44 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (12.8) | 37.9 (11.8) | 42.2 (11.1) | 38.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 13 | 47
  Male | 27 | 24 | 31 | 82
Knowledge about hearing conservation [Mean (Standard Deviation); unit: percent of correct answers] — Knowledge about hearing conservation was assessed with 16 items in the the Knowledge, Attitudes, and Behaviors Questionnaire (KAB; Saunders et al., 2014). It is a validated questionnaire that assesses knowledge about and attitudes toward hearing and hearing loss prevention. The Knowledge scale is scored as a percent correct, with a higher score indicating more knowledge.
  percent of correct answers | 57.1 (16.2) | 55.1 (16.3) | 56.7 (14.8) | 56.3 (15.7)
Susceptibility score [Mean (Standard Deviation); unit: units on a scale -50 to +50] — Perceived Susceptibility is a construct from the Health Belief Model defined as an individual's assessment of the risk of acquiring a condition. Here it assesses the extent to which the individual feels vulnerable to hearing loss. Perceived Susceptibility was assessed with 5 items in the Knowledge, Attitudes, and Behaviors Questionnaire. Scores range from -50 to +50. A higher score indicates greater perceived susceptibility.
  units on a scale -50 to +50 | 26.7 (8.8) | 29.2 (5.8) | 30.5 (6.2) | 28.8 (7.2)
Severity score [Mean (Standard Deviation); unit: units on a scale -50 to +50] — Perceived Severity is a construct from the Health Belief Model defined as an individual's assessment of the seriousness of a condition. Here it assesses the extent to which the individual believes that a hearing loss would have negative consequences. Perceived Severity was assessed with 3 items in the Knowledge, Attitudes, and Behaviors Questionnaire. Scores range from -50 to +50. A higher score indicates greater perceived severity.
  units on a scale -50 to +50 | 30.0 (19.4) | 33.3 (16.6) | 32.8 (14.0) | 32.0 (16.7)
Benefits score [Mean (Standard Deviation); unit: Units on scale -50 to +50] — Perceived Benefit is a construct from the Health Belief Model defined as an individual's assessment of the positive consequences of adopting a health behavior. Here that is the belief that hearing well is important. Perceived Benefit was assessed with 7 items in the Knowledge, Attitudes, and Behaviors Questionnaire. Scores range from -50 to +50. A higher score indicates greater perceived benefit.
  Units on scale -50 to +50 | 39.4 (12.7) | 41.4 (9.3) | 42.3 (8.7) | 41.0 (10.4)
Barriers score [Mean (Standard Deviation); unit: Units on a scale -50 to +50] — Perceived Barriers is a Health Belief Model construct defined as an individual's assessment of the influences that discourage adoption of a health behavior. Here it assesses the extent to which the individual perceives protecting hearing to be negative. Perceived Barriers was assessed with 3 items in the Knowledge, Attitudes, and Behaviors Questionnaire. Scores range from -50 to +50. A higher score indicates fewer perceived barriers.
  Units on a scale -50 to +50 | 16.1 (22.7) | 15.5 (24.1) | 15.2 (26.2) | 15.6 (24.2)
Self-efficacy score [Mean (Standard Deviation); unit: Units on a scale -50 to +50] — Perceived Self-efficacy is a Health Belief Model construct defined as an individual's assessment of their ability to successfully adopt a health behavior. Here it is the extent to which the individual believes they have the capacity to their protect hearing. It was assessed with 4 items in the Knowledge, Attitudes, and Behaviors Questionnaire. Scores range from -50 to +50. A higher score indicates greater perceived self-efficacy.
  Units on a scale -50 to +50 | 13.7 (23.3) | 9.4 (22.9) | 9.6 (23.6) | 10.9 (23.2)
Cues to action score [Mean (Standard Deviation); unit: Units on a scale -50 to +50] — Cues to action is a Health Belief Model construct defined as external influences that promote a health behavior (e.g. symptoms, media communications, or information from a healthcare provider). Here it refers to prompts from others about protecting hearing. Cues to action was assessed with 2 items in the Knowledge, Attitudes, and Behaviors Questionnaire. Scores range from -50 to +50. A higher score indicates more cues to action.
  Units on a scale -50 to +50 | 17.1 (28.4) | 20.5 (27.7) | 26.4 (24.1) | 21.4 (26.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Spent at Sound Levels >80 Decibels
Description: Objective measure of noise exposure using dosimeter to measure the percentage of time over 7days spent in sound levels >80 decibels
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Multimedia Hearing Loss Prevention Program | Hearing Conservation Brochure | Standard-of-Care
Number analyzed (Participants) | 43 | 42 | 44
percentage of time | 4.4 (0.05) | 5.0 (0.05) | 6.3 (0.06)
Statistical Analysis 1: Comparison: Multimedia Hearing Loss Prevention Program vs Hearing Conservation Brochure vs Standard-of-Care; Test type: Superiority or Other; p = 0.289, Chi-squared

2. Secondary Outcome: Knowledge About Hearing Conservation Scale
Description: Knowledge about hearing conservation was assessed with 16 items in the the Knowledge, Attitudes, and Behaviors Questionnaire (KAB; Saunders et al., 2014). It is a validated questionnaire that assesses knowledge about and attitudes toward hearing and hearing loss prevention. The Knowledge scale is scored as a percent correct, with a higher score indicating more knowledge. Data presented are for change in knowledge between baseline and 1-month follow-up computed such that a higher score indicates greater increase in knowledge.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: percent of correct answers
Groups:
- Standard-of-Care: Standard-of-Care (SoC): SoC amounts to no intervention but participants are allowed to seek information about hearing loss prevention of they want to.
Arm/Group | Multimedia Hearing Loss Prevention Program | Hearing Conservation Brochure | Standard-of-Care
Number analyzed (Participants) | 43 | 42 | 44
percent of correct answers | 11.5 (16.6) | 15.0 (14.1) | 4.7 (12.1)
Statistical Analysis 1: Comparison: Multimedia Hearing Loss Prevention Program vs Hearing Conservation Brochure vs Standard-of-Care; Test type: Superiority or Other; p = 0.004, ANOVA

3. Secondary Outcome: Change in Perceived Susceptibility Score
Description: Perceived Susceptibility is a construct from the Health Belief Model defined as an individual's assessment of the risk of acquiring a condition. In the current study it assesses the extent to which the individual feels vulnerable to hearing loss. Perceived Susceptibility was assessed with 5 items in the Knowledge, Attitudes, and Behaviors Questionnaire (KAB; Saunders et al., 2014). Scores for each item are averaged and transformed onto a scale ranging from -50 to +50, with a higher score indicating greater perceived susceptibility, which according to the Health Belief Model will increase an individual's likelihood of engaging in a health behavior. Change in Perceived Susceptibility was computed as the difference between baseline and 1-month follow-up scores, with a higher score indicating greater perceived susceptibility at follow-up.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Standard of Care: Standard of care (SoC): SoC amounts to no intervention, however protocol allows participants to independently seek information about hearing loss prevention if they want to.
Arm/Group | Multimedia Hearing Loss Prevention Program | Hearing Conservation Brochure | Standard of Care
Number analyzed (Participants) | 43 | 42 | 44
Units on a scale | 1.2 (7.9) | 0.4 (5.6) | -2.0 (6.5)
Statistical Analysis 1: Comparison: Multimedia Hearing Loss Prevention Program vs Hearing Conservation Brochure vs Standard of Care; Test type: Superiority or Other; p = 0.072, ANOVA

4. Secondary Outcome: Change in Perceived Severity Score
Description: Perceived Severity is a construct from the Health Belief Model defined as an individual's assessment of the seriousness of the consequences of a condition if it is acquired. In the current study it assesses the extent to which the individual believes that a hearing loss would have negative consequences. Perceived Severity was assessed with 3 items in the Knowledge, Attitudes, and Behaviors Questionnaire (KAB; Saunders et al., 2014). Scores for each item are averaged and transformed onto a scale ranging from -50 to +50, with a higher score indicating greater perceived severity, which according to the Health Belief Model, will increase an individual's likelihood of engaging in a health behavior. Change in Perceived Severity was computed as the difference between baseline and 1-month follow-up scores, with a higher score indicating greater perceived severity at follow-up.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Multimedia Hearing Loss Prevention Program | Hearing Conservation Brochure | Standard-of-Care
Number analyzed (Participants) | 43 | 42 | 44
Units on a scale | 7.2 (17.2) | 3.5 (13.5) | -1.7 (15.5)
Statistical Analysis 1: Comparison: Multimedia Hearing Loss Prevention Program vs Hearing Conservation Brochure vs Standard-of-Care; Test type: Superiority or Other; p = 0.030, ANOVA

5. Secondary Outcome: Change in Perceived Benefit Score
Description: Perceived Benefit is a construct from the Health Belief Model defined as an individual's assessment of the positive consequences of adopting a health behavior. In the present study that is the belief that hearing well is important. Perceived Benefit was assessed with 7 items in the Knowledge, Attitudes, and Behaviors Questionnaire (KAB; Saunders et al., 2014). Scores for each item are averaged and transformed onto a scale ranging from -50 to +50, with a higher score indicating greater perceived benefit, which according to the Health Belief Model will increase an individual's likelihood of engaging in a health behavior. Change in Perceived benefit was computed as the difference between baseline and 1-month follow-up scores, with a higher score indicating greater perceived benefit at follow-up.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Multimedia Hearing Loss Prevention Program | Hearing Conservation Brochure | Standard-of-Care
Number analyzed (Participants) | 43 | 42 | 44
units on scale | 2.6 (5.7) | .03 (8.0) | -0.8 (7.9)
Statistical Analysis 1: Comparison: Multimedia Hearing Loss Prevention Program vs Hearing Conservation Brochure vs Standard-of-Care; Test type: Superiority or Other; p = 0.092, ANOVA

6. Secondary Outcome: Change in Perceived Barriers Score
Description: Perceived Barriers is a construct from the Health Belief Model defined as an individual's assessment of the influences that discourage adoption of a health behavior. In the current study it assesses the extent to which the individual perceives few negative influences to protecting hearing. Perceived Barriers was assessed with 3 items in the Knowledge, Attitudes, and Behaviors Questionnaire (KAB; Saunders et al., 2014). Scores for each item are averaged and transformed onto a scale ranging from -50 to +50, with a higher score indicating fewer perceived barriers, which according to the Health Belief Model will increase an individual's likelihood of engaging in a health behavior. Change in Perceived Barriers was computed as the difference between baseline and 1-month follow-up scores, with a higher score indicating fewer perceived barriers at follow-up.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Multimedia Hearing Loss Prevention Program | Hearing Conservation Brochure | Standard-of-Care
Number analyzed (Participants) | 43 | 42 | 44
Units on a scale | 1.4 (14.2) | 3.2 (20.7) | 1.1 (15.2)
Statistical Analysis 1: Comparison: Multimedia Hearing Loss Prevention Program vs Hearing Conservation Brochure vs Standard-of-Care; Test type: Superiority or Other; p = 0.832, ANOVA

7. Secondary Outcome: Change in Perceived Self-efficacy Score
Description: Perceived Self-efficacy is a construct from the Health Belief Model defined as an individual's assessment of his/her ability to successfully adopt a health behavior. In the current study it assesses the extent to which the individual believes that he/she has the knowledge and abilities to protect hearing. Perceived Self-efficacy was assessed with 4 items in the Knowledge, Attitudes, and Behaviors Questionnaire (KAB; Saunders et al., 2014). Scores for each item are averaged and transformed onto a scale ranging from -50 to +50, with a higher score indicating greater perceived self-efficacy, which according to the Health Belief Model, will increase an individual's likelihood of engaging in a health behavior. Change in Perceived Self-efficacy was computed as the difference between baseline and 1-month follow-up scores, with a higher score indicating greater perceived self-efficacy at follow-up.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Multimedia Hearing Loss Prevention Program | Hearing Conservation Brochure | Standard-of-Care
Number analyzed (Participants) | 43 | 42 | 44
Units on a scale | -.2 (18.0) | -1.3 (15.3) | 3.4 (20.8)
Statistical Analysis 1: Comparison: Multimedia Hearing Loss Prevention Program vs Hearing Conservation Brochure vs Standard-of-Care; Test type: Superiority or Other; p = 0.454, ANOVA

8. Secondary Outcome: Change in Cues to Action Score
Description: Cues to action is a construct from the Health Belief Model defined as external influences that promote a health behavior (e.g. symptoms, media communications, or information from a healthcare provider). In the current study it refers to prompts from others about protecting hearing. Cues to action was assessed with 2 items in the Knowledge, Attitudes, and Behaviors Questionnaire (KAB; Saunders et al., 2014). Scores for each item are averaged and transformed onto a scale ranging from -50 to +50, with a higher score indicating greater cues to action, which according to the Health Belief Model will increase an individual's likelihood of engaging in a health behavior. Change in Cues to action was computed as the difference between baseline and 1-month follow-up scores, with a higher score indicating more Cues to action having been received at follow-up.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Multimedia Hearing Loss Prevention Program | Hearing Conservation Brochure | Standard-of-Care
Number analyzed (Participants) | 43 | 42 | 44
Units on a scale | 15.7 (24.7) | 12.8 (22.0) | 6.3 (19.3)
Statistical Analysis 1: Comparison: Multimedia Hearing Loss Prevention Program vs Hearing Conservation Brochure vs Standard-of-Care; Test type: Superiority or Other; p = 0.128, ANOVA

ADVERSE EVENTS:
Time Frame: throughout participation day 0 to study completion
Groups:
- Multimedia Hearing Loss Prevention Program: Multimedia Hearing Loss Prevention Program (HLPP) is an interactive, multimedia, computer-based HLPP that provides hands-on education and training about hearing loss, tinnitus, hearing protection, and general hearing health care for Veterans.
- Hearing Conservation Brochure: Hearing Conservation Brochure (HCB). Hearing Conservation Brochure provides knowledge-based information similar to that of the multimedia HLPP, but in written form.
- Standard of Care: Standard of Care (SoC): SoC amounts ot no intervention although participants were allowed to seek information about hearing loss prevention if they wanted to.
Arm/Group | Multimedia Hearing Loss Prevention Program | Hearing Conservation Brochure | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/44
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes